CLINICAL TRIAL: NCT05441605
Title: Effects of Chlorhexidine Solutions With Different Concentrations in Preventing Peripheral Venous Catheter-Associated Infections
Brief Title: Effect of Chlorhexidine Solution in Preventing Peripheral Venous Catheter Associated-Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Nihal Taskiran, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0000-0002-4598-6964
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Catheter-Associated Infections
Keywords: Catheter-Associated Infections; peripheral venous catheter; chlorhexidine; skin antisepsis
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Intervention Model Description: This research is a randomized controlled double-blinded experimental design. First experimental group, 1% chlorhexidine, n=24 patients, second experimental group, 2% chlorhexidine, n=24 patients, third experimental group, 4% chlorhexidine, n=24 patients, control group, 70% iso-propyl alcohol, n=24 patients
Who Masked: Participant, Investigator
Masking Description: A double-blind, experimental type of study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First group (Experimental): 1% chlorhexidine, n=24 patients.
  Interventions: Other: Effects of Chlorhexidine Solutions with Different Concentrations in Preventing Peripheral Venous Catheter-Associated Infections
- Second group (Experimental): 2% chlorhexidine, n=24 patients.
  Interventions: Other: Effects of Chlorhexidine Solutions with Different Concentrations in Preventing Peripheral Venous Catheter-Associated Infections
- Third group (Experimental): 4% chlorhexidine, n=24 patients.
  Interventions: Other: Effects of Chlorhexidine Solutions with Different Concentrations in Preventing Peripheral Venous Catheter-Associated Infections
- Fourth group (Other): control group, 70% iso-propyl alcohol, n=24 patients.
  Interventions: Other: Effects of Chlorhexidine Solutions with Different Concentrations in Preventing Peripheral Venous Catheter-Associated Infections

INTERVENTIONS:
Other: Effects of Chlorhexidine Solutions with Different Concentrations in Preventing Peripheral Venous Catheter-Associated Infections — Chlorhexidine solution in different concentrations (1%, 2%, 4%) will applied to the 3 determined experimental groups, and 70% alcohol solution will applied to the control group. Its effects in preventing peripheral venous catheter-associated infection will compared.

SUMMARY:
This research aims to determine the most effective chlorhexidine concentration to be used in preventing peripheral venous catheter-associated infections. This research is a randomized controlled double-blinded experimental design. This research will conduct between July 2022-June 2023 with 96 intensive care patients at a state hospital in Turkey. The study sample consist of 96 new insertions of peripheral venous catheters.The study will carried out as a experimental trial to compare the efficacy 1%, 2% and 4% clorhexidine gluconate and 70% alcohol in preventing infections due to catheter administrations in patients. Patients who fulfilled the inclusion criteria is randomized according to the randomization programme into three experimental groups and the control group. "Patient Information Form", "Catheter Information Form" and "Observational Form" will used to collect data.The vital findings and local infection findings of the patients that peripheral venous catheter is inserted will followed and recorded at pre-insertion and once every 24 hours for 96 hours. Culture analyze will performed from swab example taken from catheter entry location at pre-insertion,1st hour and pre removal of catheter.Data will analyzed in statistical program and p<0,05 will considered as significant.

DETAILED DESCRIPTION:
This research is a randomized controlled double-blinded experimental design. The aim of the study is to determine the most effective chlorhexidine concentration to be used in preventing peripheral venous catheter-associated infections.The study will conducted between July 2022-June 2023 at the anaesthesia and reanimation intensive care unit of a government hospital. Sample size was assessed using G-power analysis (effect size 0.3; medium level α = 0.05; 1-β = 0.80), and it was found that for each group, 24 patients had the capability of representing the population.Patients were assigned to groups using the programme random number generator.Patients who fulfilled the criteria for inclusion will taken into the study as the experimental groups (group 1: 1% chlorhexidine; group 2: 2% chlorhexidine; group 3: 4% chlorhexidine) and the control group (group 4: 70% iso-propyl alcohol).The population of the study consisted of the patients in the intensive care unit of anaesthesia and the sample consisted of the 96 adult patients who will admitted to the intensive care unit within the dates when the study was conducted and who will insertioned peripheral venous catheter and remained inpatients for at least 4 days."Patient Information Form", "Catheter Information Form" and "Observational Form" will used to collect data. The "Patient Information Form" is consisting of 13 questions about the socio-demographic information about the patient, the "Catheter Information Form" is consisting of 13 questions about the information of the catheterization, and the "Observation Form" is consisting of 13 questions about the vital findings and local infection findings of the patients. The vital findings and local infection findings of the patients that peripheral venous catheter is inserted will followed and recorded at pre-insertion and once every 24 hours for 4 days. Culture analyze will performed from swab example taken from catheter entry location at pre-insertion,1st hour and pre removal of catheter.

To perform the statistical analysis for the study, the authors will utilized the Statistical Package for Social Science (SPSS 22.0) software program. The descriptive statistics will provided in a number and percentage format. According to the Kolmogorov-Smirnov test results, key variables of the present study will analyzed using the Mann-Whitney U test for binary groups and the Kruskal-Wallis test for triple groups.and p<0,05 will considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age
* Being inpatient in the Anesthesia and Reanimation Intensive Care Unit of the hospital where the research was conducted
* No history of infection,
* No history of catheter-related infection
* No history of immunological disease
* Being an indication for peripheral venous catheter intervention

Exclusion Criteria:

* Having a central venous catheter inserted
* Having a history of allergies
* Having a history of chronic skin disease
* Peripheral venous catheter is not suitable for intervention (scar tissue in the area to be operated, wound, burn, phlebitis, infiltration, extravasation, redness, discoloration, temperature increase, tenderness, edema, drainage, pain, swelling) and in the extremity on the side of the intervention history of mastectomy, fistula, stroke)
* Presence of surgical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
H0 | one year
  Different concentrations of chlorhexidine solutions have no effect on preventing peripheral venous catheter-related infections.
  1%, 2% and 4% of chlorhexidine-gluconate solutions will compared with the 70% alcohol for skin antisepsis of PVC in ICU patients. Specimens will collected by swabbing the peripheral venous catheter entry site from the patients within before,1st and 96th hours of catheterization, respectively. The culture incubate at 37 C overnight on EMB and sheep blod agar plate. Then, the reproduction of microorganisms will identified in the culture. The presence of colonization of microorganisms in EMB blood agar indicates that gram-negative microorganism growths. The presence of colonization of microorganisms in the sheep blood agar indicates that gram-positive microorganisms growths. The absence of colonization of microorganisms in both of blood agars indicates that there is no growth.

SECONDARY OUTCOMES:
H1 | one year
  Different concentrations of chlorhexidine solutions have effect on preventing peripheral venous catheter-related infections.
  1%, 2% and 4% of chlorhexidine-gluconate solutions will compared with the 70% alcohol for skin antisepsis of PVC in ICU patients. Specimens will collected by swabbing the peripheral venous catheter entry site from the patients within before,1st and 96th hours of catheterization, respectively. The culture incubate at 37 C overnight on EMB and sheep blod agar plate. Then, the reproduction of microorganisms will identified in the culture. The presence of colonization of microorganisms in EMB blood agar indicates that gram-negative microorganism growths. The presence of colonization of microorganisms in the sheep blood agar indicates that gram-positive microorganisms growths. The absence of colonization of microorganisms in both of blood agars indicates that there is no growth.

CONTACTS AND LOCATIONS:
Overall Officials: NİHAL TAŞKIRAN, PhD, Study Director — Aydin Adnan Menderes University
Locations (1):
- TR Ministry of Health Nazilli State Hospital, Aydin, Nazi̇lli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araujo T, Rodriguez LP, Patel SA. Does my patient need a peripheral intravenous catheter? Br J Hosp Med (Lond). 2020 Jan 2;81(1):1-3. doi: 10.12968/hmed.2019.0151. Epub 2020 Jan 28. No abstract available. PMID 32003618
- [Background] Marsh N, Webster J, Mihala G, Rickard CM. Devices and dressings to secure peripheral venous catheters to prevent complications. Cochrane Database Syst Rev. 2015 Jun 12;2015(6):CD011070. doi: 10.1002/14651858.CD011070.pub2. PMID 26068958
- [Background] Alexandrou E, Ray-Barruel G, Carr PJ, Frost SA, Inwood S, Higgins N, Lin F, Alberto L, Mermel L, Rickard CM; OMG Study Group. Use of Short Peripheral Intravenous Catheters: Characteristics, Management, and Outcomes Worldwide. J Hosp Med. 2018 May 30;13(5). doi: 10.12788/jhm.3039. PMID 29813140
- [Background] Wallis MC, McGrail M, Webster J, Marsh N, Gowardman J, Playford EG, Rickard CM. Risk factors for peripheral intravenous catheter failure: a multivariate analysis of data from a randomized controlled trial. Infect Control Hosp Epidemiol. 2014 Jan;35(1):63-8. doi: 10.1086/674398. Epub 2013 Dec 2. PMID 24334800
- [Background] Keleekai NL, Schuster CA, Murray CL, King MA, Stahl BR, Labrozzi LJ, Gallucci S, LeClair MW, Glover KR. Improving Nurses' Peripheral Intravenous Catheter Insertion Knowledge, Confidence, and Skills Using a Simulation-Based Blended Learning Program: A Randomized Trial. Simul Healthc. 2016 Dec;11(6):376-384. doi: 10.1097/SIH.0000000000000186. PMID 27504890
- [Background] Macias AE, Huertas M, de Leon SP, Munoz JM, Chavez AR, Sifuentes-Osornio J, Romero C, Bobadilla M. Contamination of intravenous fluids: a continuing cause of hospital bacteremia. Am J Infect Control. 2010 Apr;38(3):217-21. doi: 10.1016/j.ajic.2009.08.015. Epub 2009 Dec 23. PMID 20031270
- [Background] Choudhury MA, Sidjabat HE, Zowawi HM, Marsh PhD N, Larsen E, Runnegar PhD N, Paterson DL, McMillan DJ, Rickard CM. Skin colonization at peripheral intravenous catheter insertion sites increases the risk of catheter colonization and infection. Am J Infect Control. 2019 Dec;47(12):1484-1488. doi: 10.1016/j.ajic.2019.06.002. Epub 2019 Jul 19. PMID 31331714
- [Background] Noorani A, Rabey N, Walsh SR, Davies RJ. Systematic review and meta-analysis of preoperative antisepsis with chlorhexidine versus povidone-iodine in clean-contaminated surgery. Br J Surg. 2010 Nov;97(11):1614-20. doi: 10.1002/bjs.7214. PMID 20878942
- [Background] Bilir A, Yelken B, Erkan A. Cholorhexidine, octenidine or povidone iodine for catheter related infections: A randomized controlled trial. J Res Med Sci. 2013 Jun;18(6):510-2. PMID 24250702
- [Background] Yamamoto N, Kimura H, Misao H, Matsumoto H, Imafuku Y, Watanabe A, Mori H, Yoshida A, Miura S, Abe Y, Toba M, Suzuki H, Ogawa K, Kanemitsu K. Efficacy of 1.0% chlorhexidine-gluconate ethanol compared with 10% povidone-iodine for long-term central venous catheter care in hematology departments: a prospective study. Am J Infect Control. 2014 May;42(5):574-6. doi: 10.1016/j.ajic.2013.12.023. Epub 2014 Mar 18. PMID 24655901
- [Background] Ohtake S, Takahashi H, Nakagawa M, Uchino Y, Miura K, Iriyama N, Nakayama T, Hatta Y, Takei M. One percent chlorhexidine-alcohol for preventing central venous catheter-related infection during intensive chemotherapy for patients with haematologic malignancies. J Infect Chemother. 2018 Jul;24(7):544-548. doi: 10.1016/j.jiac.2018.03.001. Epub 2018 Apr 4. PMID 29627326
- [Background] Capdevila JA, Guembe M, Barberan J, de Alarcon A, Bouza E, Farinas MC, Galvez J, Goenaga MA, Gutierrez F, Kestler M, Llinares P, Miro JM, Montejo M, Munoz P, Rodriguez-Creixems M, Sousa D, Cuenca J, Mestres CA; on behalf the SEICAV, SEMI, SEQ and SECTCV Societies. 2016 Expert consensus document on prevention, diagnosis and treatment of short-term peripheral venous catheter-related infections in adult. Rev Esp Quimioter. 2016 Aug;29(4):230-8. Epub 2016 Aug 28. PMID 27580009